CLINICAL TRIAL: NCT01402492
Title: Cocaine Use Reduction With Buprenorphine (CURB)
Brief Title: Cocaine Use Reduction With Buprenorphine
Acronym: CURB
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CTN-0048; U10DA013045 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Results first posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-06

CONDITIONS: Cocaine Dependence
Keywords: Cocaine-Related disorders; Cocaine; Substance-Related disorders; Opioid abuse; Opioid dependence; abuse; addiction; treatment; buprenorphine; naltrexone; Suboxone; Vivitrol
MeSH Terms: conditions — Cocaine-Related Disorders; Substance-Related Disorders; Opioid-Related Disorders; Behavior, Addictive | interventions — Buprenorphine; Naltrexone; Buprenorphine, Naloxone Drug Combination; vivitrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BUP4+XR-NTX (Experimental): 4mg buprenorphine plus naltrexone for 8 weeks of treatment
  Interventions: Drug: Buprenorphine + Naltrexone
- BUP16+XR-NTX (Experimental): 16mg buprenorphine plus naltrexone for 8 weeks of treatment
  Interventions: Drug: Buprenorphine + Naltrexone
- PLB+XR-NTX (Active Comparator): naltrexone for 8 weeks of treatment
  Interventions: Drug: Placebo + Naltrexone

INTERVENTIONS:
Drug: Buprenorphine + Naltrexone — Following a successful naloxone challenge, induction onto extended-release naltrexone by injection (Vivitrol®), and a final assessment of eligibility, participants will be randomly assigned to one of the three conditions: 4mg buprenorphine plus naltrexone, 16 mg buprenorphine plus naltrexone, or placebo plus naltrexone for 8 weeks of treatment. Random assignment will be on a 1:1:1 ratio to one of three conditions. Randomization will be stratified according to site and opioid use levels.
  Other Names: Suboxone; buprenorphine/naloxone; Vivitrol; extended release injectable naltrexone
  Arms: BUP16+XR-NTX; BUP4+XR-NTX
Drug: Placebo + Naltrexone — Following a successful naloxone challenge, induction onto extended-release naltrexone by injection (Vivitrol®), and a final assessment of eligibility, participants will be randomly assigned to one of the three conditions: 4mg buprenorphine plus naltrexone, 16 mg buprenorphine plus naltrexone, or placebo plus naltrexone for 8 weeks of treatment. Random assignment will be on a 1:1:1 ratio to one of three conditions. Randomization will be stratified according to site and opioid use levels.
  Other Names: Vivitrol; extended release injectable naltrexone
  Arms: PLB+XR-NTX

SUMMARY:
The aim of this study is to investigate the safety and effectiveness of buprenorphine in the presence of naltrexone for the treatment of cocaine dependence.

DETAILED DESCRIPTION:
This project will assess the utility of buprenorphine in the presence of naltrexone as a potential medication useful in reducing cocaine use, commencing a research direction of great importance to both theoretical and practical addiction medicine. Buprenorphine will be provided as sublingual buprenorphine+naloxone tablets (Suboxone®, "BUP"). Naltrexone will be provided as extended-release (XR) naltrexone by injection (Vivitrol®, "XR-NTX").

In this multi-center, double-blind, placebo-controlled trial, participants will randomly assigned to one of three medication conditions: 4mg buprenorphine plus naltrexone (BUP4+XR-NTX), 16mg buprenorphine plus naltrexone (BUP16+XR-NTX), or placebo plus naltrexone (PLB+XR-NTX) for 8 weeks of treatment. Participants will be scheduled for clinic visits three times weekly (for a total of 24 visits across the 8-week treatment period) for observed medication administration, provision of take-home medication, collection of safety, medical, drug use, psychological, and compliance measures. In addition, all participants will be scheduled for once-weekly individual Cognitive Behavioral Therapy (CBT) sessions.

This protocol will explore the effects of these three medication conditions to test buprenorphine as a possible treatment for cocaine dependence. This study will advance the science, provide dosing information, and characterize the effects of the combination of the two medications in this population.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years of age
* In good general health
* Meet Diagnostic and Statistical Manual (DSM)-IV criteria for cocaine dependence
* Meet DSM-IV criteria for past-year opioid dependence OR past-year opioid abuse OR have past-year opioid use and a history of opioid dependence during the lifetime
* Interested in receiving treatment for cocaine dependence
* Able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study
* Able to satisfy and comply with study procedures and requirements
* If female of childbearing potential, willing to practice and effective method of birth control for the duration of the study

Exclusion Criteria:

* Pregnant or breastfeeding females
* Known allergy or sensitivity to study medications
* Recent or ongoing treatment with medications that, in the judgment of the study medical clinician, could interact adversely with study drugs or interfere with study participation
* Have a current pattern of alcohol, benzodiazepine, or other sedative-hypnotic use, as determined by the study medical clinician, which would preclude safe participation
* Liver function test results greater than 5 times the upper limit of normal or other exclusionary clinical lab test values
* Serious medical condition or acute psychiatric disorder that would make study participation difficult or unsafe
* Pending action or situation that might prevent remaining in the area for the duration of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — University of California, Los Angeles; Andrew J. Saxon, M.D., Principal Investigator — VA Puget Sound Health Care System; Larissa J. Mooney, M.D., Principal Investigator — University of California, Los Angeles
Locations (11):
- United States (11):
  - UCLA Integrated Substance Abuse Programs (ISAP), Los Angeles, California
  - Bay Area Addiction Research and Treatment (BAART), San Francisco, California
  - Addiction Research and Treatment Services (ARTS), Denver, Colorado
  - Howard University Hospital, Washington D.C., District of Columbia
  - Atlanta VA Medical Center, Atlanta, Georgia
  - Bellevue Hospital Center, New York, New York
  - Albert Einstein College of Medicine - Division of Substance Abuse, The Bronx, New York
  - Maryhaven, Columbus, Ohio
  - CODA, Inc., Portland, Oregon
  - South Texas Veterans Health Care System, San Antonio, Texas
  - Recovery Centers of King County (RCKC), Seattle, Washington

REFERENCES:
- [Result] Ling W, Hillhouse MP, Saxon AJ, Mooney LJ, Thomas CM, Ang A, Matthews AG, Hasson A, Annon J, Sparenborg S, Liu DS, McCormack J, Church S, Swafford W, Drexler K, Schuman C, Ross S, Wiest K, Korthuis PT, Lawson W, Brigham GS, Knox PC, Dawes M, Rotrosen J. Buprenorphine + naloxone plus naltrexone for the treatment of cocaine dependence: the Cocaine Use Reduction with Buprenorphine (CURB) study. Addiction. 2016 Aug;111(8):1416-27. doi: 10.1111/add.13375. Epub 2016 Apr 21. PMID 26948856
- [Derived] Mooney LJ, Nielsen S, Saxon A, Hillhouse M, Thomas C, Hasson A, Stablein D, McCormack J, Lindblad R, Ling W. Cocaine use reduction with buprenorphine (CURB): rationale, design, and methodology. Contemp Clin Trials. 2013 Mar;34(2):196-204. doi: 10.1016/j.cct.2012.11.002. Epub 2012 Nov 16. PMID 23159524
- See also: National Institute on Drug Abuse Clinical Trials Network Website — http://www.drugabuse.gov/CTN/
- See also: Clinical Trials Network Dissemination Library Website — http://ctndisseminationlibrary.org/
- See also: UCLA Integrated Substance Abuse Programs Website — http://www.uclaisap.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- PLB+XR-NTX: Placebo plus naltrexone for 8 weeks of treatment
Period: Overall Study
Arm/Group | BUP4+XR-NTX | BUP16+XR-NTX | PLB+XR-NTX
Started | 100 | 100 | 102
Completed | 79 | 83 | 86
Not Completed | 21 | 17 | 16
Not completed — Withdrawal by Subject | 17 | 11 | 11
Not completed — Adverse Event | 2 | 3 | 4
Not completed — Physician Decision | 0 | 3 | 0
Not completed — Incarcerated (N=3) | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BUP4+XR-NTX | BUP16+XR-NTX | PLB+XR-NTX | Total
Number analyzed (Participants) | 100 | 100 | 102 | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 100 | 100 | 102 | 302
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.8 (8.00) | 45.8 (10.08) | 46.5 (7.68) | 46.3 (8.63)
Age, Customized [Number; unit: years]
  18-24 | 0 | 3 | 0 | 3
  25-34 | 9 | 14 | 7 | 30
  35-44 | 27 | 19 | 26 | 72
  45-54 | 46 | 45 | 55 | 146
  55-64 | 18 | 19 | 14 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 23 | 65
  Male | 80 | 78 | 79 | 237
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 8 | 11 | 31
  Not Hispanic or Latino | 88 | 92 | 91 | 271
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2 | 4
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 58 | 68 | 65 | 191
  White | 26 | 25 | 27 | 78
  More than one race | 5 | 5 | 6 | 16
  Unknown or Not Reported | 8 | 2 | 2 | 12
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 102 | 302

OUTCOME MEASURES:

1. Primary Outcome: Cocaine Use Days as Measured by Self-report, Corroborated by Thrice-weekly Urine Drug Screens
Description: Self-reported days of cocaine use corroborated with urine drug screens (UDS).
Time Frame: final 30 days of Treatment Phase, study days 25-54
Measure: Mean (Standard Deviation); unit: days of cocaine use
Arm/Group | BUP4+XR-NTX | BUP16+XR-NTX | PLB+XR-NTX
Number analyzed (Participants) | 100 | 100 | 102
days of cocaine use | 6.6 (5.25) | 7.2 (6.77) | 7.7 (6.16)

ADVERSE EVENTS:
Arm/Group | BUP4+XR-NTX | BUP16+XR-NTX | PLB+XR-NTX
Serious Adverse Events (participants affected / at risk) | 13/100 | 8/100 | 12/102
Other Adverse Events (participants affected / at risk) | 66/100 | 64/100 | 61/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BUP4+XR-NTX (N=100) | BUP16+XR-NTX (N=100) | PLB+XR-NTX (N=102)
Depression (Psychiatric disorders) | 1 | 1 | 0
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1
Suicidal Behavior (Psychiatric disorders) | 0 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 0
Major Depression (Psychiatric disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Drug Detoxification (Surgical and medical procedures) | 2 | 1 | 1
Dialysis (Surgical and medical procedures) | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Chest Pain (General disorders) | 2 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0 | 0
Cardiac Death (General disorders) | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BUP4+XR-NTX (N=100) | BUP16+XR-NTX (N=100) | PLB+XR-NTX (N=102)
Nausea (Gastrointestinal disorders) | 28 | 32 | 21
Vomiting (Gastrointestinal disorders) | 12 | 15 | 8
Constipation (Gastrointestinal disorders) | 10 | 10 | 9
Diarrhea (Gastrointestinal disorders) | 3 | 9 | 8
Dry Mouth (Gastrointestinal disorders) | 0 | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 1
Toothache (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 2 | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 2 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 1
Sensitivity of Teeth (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 1 | 0
Peptic Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastric Ulcer Perforation (Gastrointestinal disorders) | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Faeces Hard (Gastrointestinal disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 10 | 9 | 4
Headache (Nervous system disorders) | 9 | 6 | 5
Somnolence (Nervous system disorders) | 3 | 4 | 4
Tremor (Nervous system disorders) | 1 | 1 | 1
Sedation (Nervous system disorders) | 0 | 2 | 1
Loss of Consciousness (Nervous system disorders) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Depressed Level of Consciousness (Nervous system disorders) | 0 | 1 | 0
Tension Headache (Nervous system disorders) | 1 | 0 | 0
Aura (Nervous system disorders) | 0 | 0 | 1
Parosmia (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 5 | 2
Depression (Psychiatric disorders) | 3 | 2 | 2
Anxiety (Psychiatric disorders) | 1 | 5 | 0
Libido Decreased (Psychiatric disorders) | 2 | 0 | 3
Suicidal Ideation (Psychiatric disorders) | 0 | 3 | 2
Euphoric Mood (Psychiatric disorders) | 1 | 1 | 0
Depressed Mood (Psychiatric disorders) | 1 | 0 | 1
Sleep Disorder (Psychiatric disorders) | 1 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 1 | 0
Intentional Self-injury (Psychiatric disorders) | 0 | 1 | 0
Drug Dependence (Psychiatric disorders) | 0 | 0 | 1
Disorentation (Psychiatric disorders) | 0 | 1 | 0
Suicidal Behavior (Psychiatric disorders) | 0 | 0 | 1
Substance-induced Mood Disorder (Psychiatric disorders) | 0 | 1 | 0
Psychotic Disorder (Psychiatric disorders) | 1 | 0 | 0
Panic Attack (Psychiatric disorders) | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1
Major Depression (Psychiatric disorders) | 0 | 1 | 0
Fatigue (General disorders) | 9 | 6 | 4
Drug Withdrawal Syndrome (General disorders) | 2 | 2 | 3
Irritability (General disorders) | 3 | 0 | 0
Chest Pain (General disorders) | 2 | 0 | 1
Non-cardiac Chest Pain (General disorders) | 2 | 0 | 0
Influenza-like Illness (General disorders) | 0 | 2 | 0
Sluggishness (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Limb Discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 3
Tooth Abscess (Infections and infestations) | 0 | 3 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 2
Tooth Infection (Infections and infestations) | 0 | 1 | 0
Periorbital Infection (Infections and infestations) | 0 | 0 | 1
Haemophilus Infection (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 5 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Cold Sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Acute Febrile Neutrophilic Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Astma (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Decreased Appetitie (Metabolism and nutrition disorders) | 4 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 2
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-traumatic Neck Syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post-lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Drug Detoxification (Surgical and medical procedures) | 2 | 1 | 1
Tooth Extraction (Surgical and medical procedures) | 0 | 1 | 0
Dialysis (Surgical and medical procedures) | 0 | 1 | 0
Weight Increased (Investigations) | 1 | 0 | 0
Urine Analysis Abnormal (Investigations) | 0 | 1 | 0
Liver Function Test Abnormal (Investigations) | 1 | 0 | 0
International Normalized Ratio Increased (Investigations) | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 0 | 1 | 0
Hot Flush (Vascular disorders) | 1 | 1 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to Spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seasonal Allergy (Immune system disorders) | 2 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0
Ear Discomfort (Ear and labyrinth disorders) | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Lacrimation Increased (Eye disorders) | 1 | 0 | 0
Hyperthyrodism (Endocrine disorders) | 1 | 0 | 0
Adrenal Mass (Endocrine disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Monocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results. The sponsor can require changes to the communication and can extend the embargo.